CLINICAL TRIAL: NCT01311141
Title: Target Site Pharmacokinetics of Doripenem After a Single Dose of 500mg in Healthy Volunteers - a Pilot Study
Brief Title: Target Site Pharmacokinetics of Doripenem After a Single Dose of 500mg in Healthy Volunteers Dori_MD_1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2010-020778-41
Record Dates: First submitted 2011-03-08; First posted 2011-03-09 (Estimated); Last update posted 2011-04-01 (Estimated); Status verified 2010-08

CONDITIONS: Healthy
MeSH Terms: interventions — Doripenem

ARMS (1):
- Doripenem i.v. (Experimental): no comparator, PK study
  Interventions: Drug: doripenem

INTERVENTIONS:
Drug: doripenem — doripenem once i.v.500mg

SUMMARY:
In the present study we will measure and compare the unbound, i.e. microbiologically active concentrations of doripenem after a single dose of 500mg in plasma, subcutaneous adipose tissue and muscle tissue and saliva of healthy volunteers. We will use the microdialysis technique, which allows for the continuous measurement of unbound drug concentrations in the interstitial space fluid. The findings of the present study will help to assess whether currently employed therapy regimens with doripenem provide effective antimicrobial concentrations in different compartments in man

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Male

Exclusion Criteria:

* Female
* Ill

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2010-08; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
The time versus unbound doripenem concentration profiles in the interstitial space fluid of non inflamed subcutaneous adipose tissue, muscle tissue, saliva and plasma

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria